CLINICAL TRIAL: NCT00821509
Title: STOPFLU: Is it Possible to Reduce the Number of Days Off in Office Work by Improved Hand-hygiene?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Finnish Work Environment Fund (Other); Finnish Institute of Occupational Health (Other); Berner Oy (Industry); Farmos Oy (Industry); Kesko Oyj (Unknown); Nordea Bank Finland Plc (Unknown); Outokumpu (Unknown); Outokumpu Technogy Oyj (Unknown); Suomen Osuuskauppojen Keskuskunta (SOK) (Unknown); S-Pankki (Other)
Responsible Party: Principal Investigator, Tapani Hovi, Project Leader, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: KTL460-8
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Results first posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-02

CONDITIONS: Respiratory Infection; Gastroenteritis
Keywords: virus infection; hygiene; transmission; intervention
MeSH Terms: conditions — Respiratory Tract Infections; Gastroenteritis; Virus Diseases | interventions — Hand Disinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hand washing (Active Comparator): Instructions for proper coughing and sneezing, and for reduced hand shaking; frequent hand washing in office and at home
  Interventions: Behavioral: Hand washing
- Disinfectant rubbing (Active Comparator): Instructions for proper coughing and sneezing, and for reduced hand shaking; frequent rubbing of hands with alcohol containing disinfectant in office and at home
  Interventions: Behavioral: Disinfectant rubbing
- Control (No Intervention): No change in hygiene behaviour

INTERVENTIONS:
Behavioral: Hand washing — Instructions for proper coughing and sneezing, and for reduced hand shaking, frequent hand washing in office and at home
  Arms: Hand washing
Behavioral: Disinfectant rubbing — Instructions for proper coughing and sneezing, and for reduced hand shaking; frequent rubbing of hands with alcohol containing disinfectant in office and at home
  Arms: Disinfectant rubbing

SUMMARY:
Improved hand hygiene is known to reduce transmission of both respiratory (RTI) and gastrointestinal infections (GTI) under "semi-closed" conditions such as hospitals, day-care centres and schools. It is not known if similar interventions would have the desired effect in a regular office work. This study is aiming to investigate this possibility by recruiting volunteers from several companies in the Helsinki Region. The two intervention groups will receive detailed instructions e.g. for proper coughing and sneezing, and for regular cleaning of hands with either standard liquid soap or with alcohol-based gel rubbing. Third group will serve as the control and is advised not to change their previous behaviour in this respect. The participants will report weekly possible RTI or GTI symptoms and related days off through internet. The study is planned to run about 18 months to cover the seasonal variation of the epidemics of the causative different viruses.

DETAILED DESCRIPTION:
It is common knowledge that both respiratory tract infections (RTI) and gastrointestinal infections (GTI) cause a large part of short periods of days off from work, day care and school. In addition, because of the generally mild nature of the diseases, especially adults often come to work in spite of symptoms, and may therefore initiate transmission of infection among their colleagues. The chain of events from exposure to a pathogenic virus to subsequent infection and staying home because of infectious disease is a very complicated one, and is affected by many factors potentially causing variation, such as the multitude of causative agents, different individual histories of infections, variability of inter-personal contacts in work and various working- team feelings -influenced thresholds for staying home etc. Therefore, we aim to recruit at least 24 operationally distinct volunteer groups, each including at least 50 persons, and to continue the intervention about 18 months.

A virus transmission "risk-index" will be calculated for each group based on potential participant questionnaires enquiring, among other things, about numbers and ages of children, their possible out-of-home day care, personal properties such as smoking, chronic diseases, and potential differences in contacts during daily work. The 24 groups will be divided in groups of three most similar ones, and members each triplet then randomised in one the intervention groups or the control (see brief summary).

Data collection is based on self-reporting through Monday-morning electronic reports using a standard form. The from is enquiring about possible exposure to persons suffering from RTI or GTI, and possible own symptoms of the same diseases during the preceding 7 day period (including weekends and other holidays). The form will require daily records offering all possible combinations of the following categories: healthy-with symptoms, working normally-day off, own disease-child ill-other reason for day off.

Etiology of the symptoms will not be searched for on individual basis in this study but a connection to RTI virus epidemiology is built by a sentinel surveillance, where occupational health clinics located in the premises of the participating companies send a standard number of weekly specimens collected from employees visiting the clinic. For possible GTI outbreaks a standard outbreak investigation principle will be followed, including 3-5 specimens. from typical patients will be collected. Common causative agents of the diseases will be searched for using real-time PCR techniques.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers working in defined units

Exclusion Criteria:

* Persons with open wounds or chronic eczema in hands

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tapani Hovi, MD PhD, Study Director — National Public Health Institute, Finland
Locations (1):
- National Institute for Health and Wellfare (THL), Helsinki, Finland

REFERENCES:
- [Derived] Jefferson T, Dooley L, Ferroni E, Al-Ansary LA, van Driel ML, Bawazeer GA, Jones MA, Hoffmann TC, Clark J, Beller EM, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2023 Jan 30;1(1):CD006207. doi: 10.1002/14651858.CD006207.pub6. PMID 36715243
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Hovi T, Ollgren J, Savolainen-Kopra C. Intensified hand-hygiene campaign including soap-and-water wash may prevent acute infections in office workers, as shown by a recognized-exposure -adjusted analysis of a randomized trial. BMC Infect Dis. 2017 Jan 9;17(1):47. doi: 10.1186/s12879-016-2157-z. PMID 28068912
- [Derived] Hovi T, Ollgren J, Haapakoski J, Savolainen-Kopra C. Development of a prognostic model based on demographic, environmental and lifestyle information for predicting incidences of symptomatic respiratory or gastrointestinal infection in adult office workers. Trials. 2016 Nov 16;17(1):545. doi: 10.1186/s13063-016-1668-7. PMID 27852324
- [Derived] Hovi T, Ollgren J, Haapakoski J, Amiryousefi A, Savolainen-Kopra C. Exposure to persons with symptoms of respiratory or gastrointestinal infection and relative risk of disease: self-reported observations by controls in a randomized intervention trial. Trials. 2015 Apr 17;16:168. doi: 10.1186/s13063-015-0691-4. PMID 25879224
- [Derived] Savolainen-Kopra C, Haapakoski J, Peltola PA, Ziegler T, Korpela T, Anttila P, Amiryousefi A, Huovinen P, Huvinen M, Noronen H, Riikkala P, Roivainen M, Ruutu P, Teirila J, Vartiainen E, Hovi T. STOPFLU: is it possible to reduce the number of days off in office work by improved hand-hygiene? Trials. 2010 Jun 4;11:69. doi: 10.1186/1745-6215-11-69. PMID 20525328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Occupational health clinics of 6 corporations in the Helsinki region contacted in 2008; 21 study clusters identified with at least. 50 employees in common office work in each; Active recruitment by personal invitation to all members of the identified clusters (N=1270)in early January 2009 by emails including a designated risk interview (see below)
Pre-assignment Details: Based on the cumulated acute infection risk (day-care of children, age, smoking, chronic CV- or lung disease, frequent business travel etc.)in each cluster the clusters were ranked according to the calculated risk index, and out of the 7 cluster triplets with most similar index, one was randomly allocated to each of the three study arms
Period: Overall Study
Arm/Group | Hand Washing | Disinfectant Rubbing | Control
Started | 257 | 202 | 224
Completed | 245 (This is a result of 56 lost-to-follow-up and 44 new recruits) | 191 (This is a result of 57 lost-to-follow-up and 46 new recruits) | 190 (This is a result of 50 lost-to-follow-up and 16 new recruits)
Not Completed | 12 | 11 | 34
Not completed — Withdrawal by Subject | 12 | 11 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hand Washing | Disinfectant Rubbing | Control | Total
Number analyzed (Participants) | 257 | 202 | 224 | 683
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 257 | 202 | 224 | 683
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 153 | 163 | 501
  Male | 72 | 49 | 61 | 182
Region of Enrollment [Number; unit: participants]
  Finland | 257 | 202 | 224 | 683

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Reported Days-off Episodes in the Arm Due to Own Infectious Disease Over the Total Number of Follow-up Weeks in the Arm
Description: Participants reported weekly through an internet questionnaire symptoms of respiratory tract (RTI) or gastrointestinal tract infections (GTI) as well as whether they were working (if expected) or not, daily for the previous calendar week. Individual weekly reports were combined in a single continuum and successive days with both symptoms and absence from work were designated as days-off episodes due to own infectious disease. Number of these episodes in each trial arm was calculated and for the respective proportion, was divided by the total number of weekly reports collected in the arm.
Time Frame: At the end of the entire study period (16 months)
Population: Number of participants given is the number at the onset. There were both lost-to-follow-up and new recruits. The analysis is, however, based on episodes of days-off in entire arm during the entire follow-up time rather than on individual participants
Measure: Number; unit: sick-leave episodes
Units Other Than Participants: Reported follow-up weeks
Groups:
- Hand Washing: Participants received behavioural instructions how to limit transmission of infections and were recommended to wash hand frequently
- Disinfectant Rubbing: Participants received behavioural instructions how to limit transmission of infections and were recommended to clean their hands frequently with an alcohol containing disinfectant solution
- Control: Participants were advised not to change their hand hygiene habits
Arm/Group | Hand Washing | Disinfectant Rubbing | Control
Number analyzed (Participants) | 257 | 202 | 224
Number analyzed (Reported follow-up weeks) | 15014 | 11986 | 11644
sick-leave episodes | 625 | 418 | 405
Statistical Analysis 1: Comparison: Hand Washing vs Control; According to the null hypothesis the proportion of weeks with an onset of days-off period in neither of the intervention arms was different from that of control. No in advance power calculations were done; Test type: Superiority or Other; p = 0.004, proportion test; The test was carried out using the proportions calculated from the number of sick-leave episodes over the number o total follow-up weeks in each arm; ratio of proportions = 1.03

2. Primary Outcome: Cumulative Number of Reported Episodes of Infectious Disease in the Arm Over the Total Number of Follow-up Weeks in the Arm
Description: Participants reported weekly through an internet questionnaire symptoms of respiratory tract (RTI) or gastrointestinal tract infections (GTI). Individual weekly reports were combined in a single continuum and successive days with either RTI or GTI symptoms were designated as disease episodes due. Numbers of RTI, GTI and either episodes in each trial arm were calculated, and for the respective proportion, were divided by the total number of weekly reports collected in the arm.
Time Frame: At the end of the study period (16 months)
Population: as for outcome 1
Measure: Number; unit: Disease episodes
Units Other Than Participants: Follow-up weeks
Arm/Group | Hand Washing | Disinfectant Rubbing | Control
Number analyzed (Participants) | 257 | 202 | 224
Number analyzed (Follow-up weeks) | 15014 | 11986 | 11644
Disease episodes | 1451 | 1288 | 1214
Statistical Analysis 1: Comparison: Hand Washing vs Control; According to the null hypothesis the proportion of weeks with an onset of an infectious disease period in neither of the intervention arms was different from that of control. No in advance power calculations were done; Test type: Superiority or Other; p = 0.04, proportion test; ratio of proportions = 0.933

ADVERSE EVENTS:
Time Frame: Entire follow up period of 16 months
Arm/Group | Hand Washing | Disinfectant Rubbing | Control
Serious Adverse Events (participants affected / at risk) | 0/257 | 0/202 | 0/224
Other Adverse Events (participants affected / at risk) | 0/257 | 0/202 | 0/224

LIMITATIONS AND CAVEATS:
In a pre-study interview, 90% stated "when I have cold I usually come to work if I only can". Participants in the intervention arms, but not those of the control arm, were advised to stay home when sick: possible contribution to outcome measure 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes